CLINICAL TRIAL: NCT01382667
Title: Evaluation of Dyspeptic Symptoms in Oncological Frail Patients With Extraintestinal Cancer in Chemotherapy. Assessment of Circulating Levels of Glucagon-like Peptide 2 (GLP-2) in Relation to Mucositis
Brief Title: Plasma Levels of Glucagon-like Peptide-2 and Dyspepsia in Patients With Extraintestinal Cancer During Chemotherapy
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Francesco Russo, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: SRLP06
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Lung Cancer; Dyspepsia
Keywords: mucositis; dyspepsia; chemotherapy; GLP-2; questionnaire
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Dyspepsia; Mucositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GLP-2 and symptom evaluation: Before starting and at the end of the chemotherapy, along with a blood withdrawal for GLP-2 evaluation, a GSRS (gastrointestinal symptom rate scale) questionnaire will be filled by each patient to account for GI symptoms. In addition, minor complaints such as warm sensation after chemotherapy, susceptibility to nausea under specific condition, sweating and weakness will scored by visual analog score (VAS). Lastly, the NCI-CTC score for mucositis will be performed.

SUMMARY:
The specific aim of the study is to investigate the relationship between the development of dyspepsia and GI dyspeptic symptoms in relation to circulating levels of peculiar GI peptides (such gastrin, pepsinogen and GLP-2) in patients with non-gastrointestinal neoplasm well controlled for emesis.

DETAILED DESCRIPTION:
The complications of anticancer treatment threaten the effectiveness of therapy because they lead to dose reduction, increase healthcare costs, and impair patients' quality of life. Gastrointestinal (GI) symptoms are the most frequent side effects of antineoplastic chemotherapy behind bone-marrow depression, with nausea and vomiting representing the mainly referred ones.

Gastrointestinal (GI) mucositis, which represents injury of the rest of the alimentary tract beyond oral mucositis, is becoming recognized increasingly as a toxicity associated with many standard-dose chemotherapy regimens. Although clinicians consider them "minor complaints", many patients (40-100%) treated with chemotherapy and/or exposed to ionizing radiation suffer from such a disease. After chemotherapy, GI mucositis is most prominent in the small intestine, but it also occurs in the esophagus, stomach, and large intestine. The GI symptoms related to mucositis mimic those from other GI disease (such as dyspepsia, reflux disease or abdominal pain and diarrhea). Alimentary tract mucositis increases morbility and mortality and contribute to rising health care cost.

The comprehension of pathophysiology will shed light on the rationale for targeting specific pathways and so for the use of specific agents for prevention and treatment. Since the role of chemotherapy in the onset of GI motility disorders in addition to minor GI complaints has not been clarified yet. Understanding the pathophysiology of mucositis, its measures and scores, are essential for progress in research and care direct at this common side-effect of anticancer therapy. Currently, there is not strong evidence to support a recommendation for and against the use of certain agents (mucosal surface protectants, antiinflammatory or antimicrobial agents, growth factors, etc).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed cancer (lung and breast cancer),
* Patients currently free of active disease

Exclusion Criteria:

* History of cerebral edema, primary and secondary brain neoplasm with signs and symptoms of raised intracranial pressure and/or brain metastases,
* Signs of marked hepatic or renal dysfunction, cardiac failure
* Signs of dyspepsia, peptic ulcer, gastric surgery or prior diagnosis of other cancer
* Administration of drugs interfering with GI motility (i.e. antisecretory, prokinetic, or antibiotic drugs) as well as the exposition to radiotherapy, four weeks prior to the examination
* Referred episode of nausea of any severity within 24 h prior to antiemetic therapy, if they had experienced vomiting in the previous 24 h,
* Pregnancy or lactating
* Concomitant administration of agents known to have significant antiemetic activity, including benzodiazepines and other corticosteroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-five patients who had undergone surgical ablation of the primitive tumour (lung and breast cancer) as definitive primary treatment and attending the Oncology Day Hospital of our Institute,and the IRCCS Oncologico of Bari will be enrolled. They had to be scheduled for adjuvant therapies associated with a standard dosage of antiserotoninergic drugs according to ESMO recommendations
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
GLP-2 plasma levels in cancer patients | 21 days
  Evaluation of plasma levels of GLP-2 in patients with extraintestinal cancer before and after chemotherapy.

SECONDARY OUTCOMES:
Cancer associated dyspepsia syndrome, mucositis and GLP-2 plasma levels | 21 days
  Evaluation of the symptom profile related to CADS (cancer associated dyspepsia syndrome) before and after the first cycle of chemotherapy.
  Assessment of possible relations between mucositis score, gastrointestinal symptom score and GLP-2 plasma levels.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Clemente, ScD, Principal Investigator — National Institute of Digestive Diseases IRCCS "S. de Bellis"
Locations (1):
- National Institute for Digestive Diseases IRCCS "S. de Bellis", Castellana Grotte, Bari, Italy

REFERENCES:
- [Background] Riezzo G, Chiloiro M, Russo F, Clemente C, Di Matteo G, Guerra V, Di Leo A. Gastric electrical activity and gastrointestinal hormones in dyspeptic patients. Digestion. 2001;63(1):20-9. doi: 10.1159/000051868. PMID 11173896
- [Background] Drucker DJ. Biological actions and therapeutic potential of the glucagon-like peptides. Gastroenterology. 2002 Feb;122(2):531-44. doi: 10.1053/gast.2002.31068. PMID 11832466
- [Background] Riezzo G, Clemente C, Leo S, Russo F. The role of electrogastrography and gastrointestinal hormones in chemotherapy-related dyspeptic symptoms. J Gastroenterol. 2005 Dec;40(12):1107-15. doi: 10.1007/s00535-005-1708-7. PMID 16378174
- [Background] Peterson DE, Cariello A. Mucosal damage: a major risk factor for severe complications after cytotoxic therapy. Semin Oncol. 2004 Jun;31(3 Suppl 8):35-44. doi: 10.1053/j.seminoncol.2004.04.006. PMID 15181607
- [Background] Hesketh PJ, Van Belle S, Aapro M, Tattersall FD, Naylor RJ, Hargreaves R, Carides AD, Evans JK, Horgan KJ. Differential involvement of neurotransmitters through the time course of cisplatin-induced emesis as revealed by therapy with specific receptor antagonists. Eur J Cancer. 2003 May;39(8):1074-80. doi: 10.1016/s0959-8049(02)00674-3. PMID 12736106
- [Derived] Russo F, Linsalata M, Clemente C, D'Attoma B, Orlando A, Campanella G, Giotta F, Riezzo G. The effects of fluorouracil, epirubicin, and cyclophosphamide (FEC60) on the intestinal barrier function and gut peptides in breast cancer patients: an observational study. BMC Cancer. 2013 Feb 4;13:56. doi: 10.1186/1471-2407-13-56. PMID 23379680